CLINICAL TRIAL: NCT01662284
Title: A Phase 1/2 Study of 124I-NM404 in Subjects With Advanced Solid Malignancies
Brief Title: Study of 124I-NM404 in Advanced Solid Malignancies
Status: Terminated | Type: Observational
Why Stopped: Sponsor determined this trial does not support their anticipated clinical development program.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CO12901; 2012-0230 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2012-01953 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2012-08-03; First posted 2012-08-10 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2017-01

CONDITIONS: Triple Negative Breast, Prostate, Colorectal, Gastric, Ovarian, Pancreatic, Esophageal, Soft Tissue Sarcoma, and Head & Neck Cancer
MeSH Terms: conditions — Sarcoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Triple Negative Breast: 124I-NM404 in triple negative breast cancer
  Interventions: Drug: 124I-NM404
- Prostate: 124I-NM404 in prostate cancer
  Interventions: Drug: 124I-NM404
- Colorectal: 124I-NM404 in colorectal cancer
  Interventions: Drug: 124I-NM404
- Gastric: 124I-NM404 in gastric cancer
  Interventions: Drug: 124I-NM404
- Ovarian: 124I-NM404 in ovarian cancer
  Interventions: Drug: 124I-NM404
- Pancreatic: 124I-NM404 in pancreatic cancer
  Interventions: Drug: 124I-NM404
- Esophageal: 124I-NM404 in esophageal cancer
  Interventions: Drug: 124I-NM404
- Sarcoma: 124I-NM404 in soft tissue sarcoma
  Interventions: Drug: 124I-NM404
- Head & Neck: 124I-NM404 in head and neck cancer
  Interventions: Drug: 124I-NM404

INTERVENTIONS:
Drug: 124I-NM404 — 124I-NM404 administered at either 5mCi or 3mCi on day 1. If PET/CT images are diagnostically inadequate and there are no dose-limiting toxicities at current dose, next patients will receive the next higher level of 7.5 or 10 mCi.

SUMMARY:
The purpose of this study is to assess the use of investigational compound 124I-NM404 for accurate detection and characterization of a wide variety of solid primary and metastatic malignancies anywhere in the body.

DETAILED DESCRIPTION:
124I-NM404 is a new investigational agent being developed to better identify local tumors and cancerous tumors using imaging technologies such as positron emission tomography (PET) scans. An investigational drug is a drug that has not been approved by the Food and Drug Administration (FDA) and is available for research use only. 124I-NM404 is only taken up by the cancer cells, not the normal cells. Compared to traditional methods such as CT (computed tomography) or MRI (Magnetic resonance imaging), 124I-NM404 may help physicians more accurately see and evaluate cancerous tumors. This agent has been safely studied in animals and a limited number of human patients with lung cancer. This study is being done to determine the best dose to use and to fully evaluate the images that result from using this new agent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced solid malignancy.
* Allowed tumor types: triple negative breast, prostate, colorectal, gastric, ovarian, pancreatic, esophageal, soft tissue sarcoma, and head & neck cancer
* Disease must be at least 1cm in diameter
* Brain metastasis must be stable for at least one month.
* ECOG performance status 0-2
* Anticipated survival less than 5 years, as per the treating physician

Exclusion Criteria:

* Skin lesions only
* Chemotherapy or radiotherapy within 1 week
* Residual toxicities of grade 2 or greater from prior therapy
* Adequate organ function as per specified laboratory parameter
* Platelet count > or = to 75,000/uL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be referred to the Phase I oncology research office by their treating oncologist. Outside referrals will be managed by Cancer Connect who will ensure that potential subjects are first evaluated by a UW medical oncologist in the cancer clinic who will then refer them, if appropriate, to the Phase I oncology office.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Optimal Imaging Parameters | 2 years
  To determine the optimal imaging parameters (dose, acquisition time, imaging time post injection, normal organ and tumor dosimetry) of 124I-NM404 in subjects with advanced solid malignancies with one of the following tumor types: triple negative breast, prostate, colorectal, gastric, ovarian, pancreatic, esophageal, soft tissue sarcoma, and head & neck cancer

SECONDARY OUTCOMES:
Adverse events | 2 years
  Number and grade of adverse events attributable to 124I-NM-404
PET comparison | 2 years
  compare 18F-FDG PET to 124I-NM404 PET

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/